CLINICAL TRIAL: NCT03610659
Title: Validity and Reliability of The Turkish Version of Assessment of Burden of COPD Scale
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Seda Saka, MSc, PT, Bezmialem Vakif University
Other Study IDs: ssaka03
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: COPD
Keywords: COPD; Burden of disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In our study, we aimed to evaluate the validity and reliability of the Turkish version of theAssessment of Burden of COPD (ABC) Scale.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common pulmonary disease characterized by airway limitation, irreversible, preventable, and treatable (1,2). COPD is a major health problem that affects the entire world and is expected to be the fourth, the seventh, cause of death in 2030 (3). The concept of "holistic assessment of disease burden" is widely used to support the personalized care management of COPD patients. Disease burden; physical, psychological, emotional and / or social burden felt by the patient. When the questionnaires in the literature evaluating the quality of life / health status in COPD patients were examined, it was seen that none of these questionnaires included all aspects of COPD burden definition (4). Clinical COPD Questionnaire (CCQ) is a 10-question questionnaire that assesses COPD burden in most aspects and situations. Assessment of Burden of COPD (ABC) Scale was developed to evaluate the burden of disease in COPD patients by adapting this questionnaire. The ABC scale was formed by combining three items (a short tool for early identification of distress) and a substance that measures fatigue with the questions of the CCQ scale. As a result, a scale of 14 items with 5 fields was formed.

ELIGIBILITY:
Inclusion Criteria:

* FEV1/FVC<%70
* To be able to read and understand Turkish

Exclusion Criteria:

* Having undergone a COPD exacerbation in the last 6 weeks
* Having comorbidities affecting ambulance
* Having cognitive disorders

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-06-23 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Burden of COPD (ABC) Scale | 3 Minutes
  The ABC scale is a 14-item newly developed COPD burden assessment questionnaire that the person responds to on their own. The scale includes questions that are objective determinants of COPD disease burden integrated with the health status of the patient. There is a total score and 5 subtitle scores; symptoms (4 items), functional status (4 items), mental condition (2 items), emotional condition (3 items) and fatigue (1 item). Scoring is done between 0 and 6 (0 = no disease burden, 6 = high disease burden).

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Slok AH, Bemelmans TC, Kotz D, van der Molen T, Kerstjens HA, In 't Veen JC, Chavannes NH, Asijee GM, Rutten-van Molken MP, van Schayck OC. The Assessment of Burden of COPD (ABC) Scale: A Reliable and Valid Questionnaire. COPD. 2016 Aug;13(4):431-8. doi: 10.3109/15412555.2015.1118025. Epub 2016 Jan 20. PMID 26788838
- [Background] Goossens LMA, Rutten-van Molken MPMH, Boland MRS, Donkers B, Jonker MF, Slok AHM, Salome PL, van Schayck OCP, In 't Veen JCCM, Stolk EA; research team that developed the ABC tool.. ABC Index: quantifying experienced burden of COPD in a discrete choice experiment and predicting costs. BMJ Open. 2017 Dec 26;7(12):e017831. doi: 10.1136/bmjopen-2017-017831. PMID 29282261